CLINICAL TRIAL: NCT06607796
Title: A Multicenter Study of the Efficacy and Safety of Intratumoral Injection of Toluenesulfonamide (PTS) in Combination With or Without First-line Chemoimmunotherapy Based on Standard Treatment for Stage IV Driver Gene-negative Non-small Cell Lung Cancer
Brief Title: Efficacy and Safety of Intratumoral Toluenesulfonamide (PTS) Injection in Stage IV Driver Gene-Negative NSCLC With/Without Chemoimmunotherapy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zhou Chengzhi (Other)
Responsible Party: Sponsor-Investigator, Zhou Chengzhi, chief physician, Guangzhou Institute of Respiratory Disease
Organization: Guangzhou Institute of Respiratory Disease (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CROC-24-09
Record Dates: First submitted 2024-09-18; First posted 2024-09-23 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — 6-pyruvoyltetrahydropterin synthase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): intratumoral injection of toluenesulfonamide (PTS) to oligo lesions
  Interventions: Drug: Toluenesulfonamide (PTS) Intratumoral Injection
- Control subjects (No Intervention): follow-up observation of oligofocal lesions, no PTS intratumoral injection treatment, if progression can be oligofocal PTS intratumoral injection

INTERVENTIONS:
Drug: Toluenesulfonamide (PTS) Intratumoral Injection — intratumoral injection of toluenesulfonamide(PTS) to oligo lesions
  Arms: Experimental group

SUMMARY:
The aim of this study was to evaluate the efficacy and safety of intratumoral injection of toluenesulfonamide(PTS) in combination with or without first-line chemoimmunization based on standard treatment for stage IV driver gene-negative non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand, be informed about the study and sign the Informed Consent Form (ICF); be willing to follow and be capable of completing all trial procedures；
2. Age ≥18 years and ≤75 years at the time of signing the ICF；
3. Histologically or cytologically confirmed stage IV (AJCC 8th edition) driver gene negative non-small cell lung cancer；
4. At least one measurable target lesion assessed by the investigator according to the requirements of RECIST 1.1 within 4 weeks prior to enrollment, except for lesions proposed for percutaneous PTS local injection；
5. Localized injectable lesions located in a more confined area of the outer lung bands, less than or equal to 5 cm in diameter; these may be primary lesions that are not amenable to surgical resection or localized recurrent lesions after surgical resection and radiotherapy treatment；
6. ECOG PS score of 0 or 1 within 7 days prior to local treatment tolerates PTS intratumoral injections；
7. Patients with localized lesions present and persistently stable (SD evaluated after two courses of treatment) after standard treatment with first-line chemoimmunotherapy；
8. Life expectancy ≥ 3 months；
9. Normal liver, kidney and heart function, normal blood routine, blood biochemistry, coagulation function and electrolytes and other physiological indicators.

Exclusion Criteria:

1. Plans for radiotherapy, surgery, etc. for the lesion after intratumor injection;
2. Have severe cardiopulmonary dysfunction, advanced hepatic or renal insufficiency, malignant cardiac arrhythmia, hypertension, etc;
3. Have severe bleeding, clotting disorders, infections, dehydration, etc;
4. Have blood disorders, autoimmune diseases, cirrhosis of the liver, etc;
5. History of severe emphysema and pulmonary alveoli;
6. History of drug allergy or contraindication to toluene sulfonamide;
7. Women who are pregnant, breastfeeding, or planning to become pregnant during the study period;
8. The investigators determined that the patients had other conditions that made them unsuitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | 3 years
  Proportion of target lesions stabilized after two courses of first-line chemoimmunotherapy standard therapy combined with and without PTS intratumoral injection, with tumor volume reduction to achieve complete remission (CR) and partial remission (PR)

SECONDARY OUTCOMES:
Median progression-free survival(mPFS) | 3 years
  Time from receipt of first-line chemoattenuated standard of care in combination with or without PTS intratumoral injection until first objectively documented disease progression or death from any cause (whichever occurs first)
Median overall survival(mOS) | 3 years
  Time from receipt of first-line chemoattenuated standard of care in combination with or without PTS intratumoral injection until death from any cause (whichever occurs first)

CONTACTS AND LOCATIONS:
Overall Officials: Chengzhi Zhou, doctor, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University,Guangzhou
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China